CLINICAL TRIAL: NCT04157647
Title: Monocentric Prospective Randomized Pilot Study in Patients With Kidney Failure to Evaluate the Relationship Between the Hemadsorption During and After Cardiopulmonary Bypass and the Modulation of Post-surgical Inflammatory Response
Brief Title: Hemadsorption During and After Cardiopulmonary Bypass to Modulate the Inflammatory Response
Acronym: IMHeS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Magna Graecia (Other)
Responsible Party: Principal Investigator, GIUSEPPE FILIBERTO SERRAINO, Principal Investigator, University Magna Graecia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: IMHeS
Record Dates: First submitted 2019-10-13; First posted 2019-11-08 (Actual); Last update posted 2020-11-12 (Actual); Status verified 2020-11

CONDITIONS: Inflammatory Response; Chronic Renal Disease; Cardiac Surgery
Keywords: hemadsorption
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CytoSorb (Active Comparator): Patients assigned to this arm group will receive hemadsorption witbhCytoSorb during the surgery and in the next 24 hours after surgery.
  Interventions: Device: CytoSorb
- Control (Sham Comparator): Patients assigned to this arm group will undergo to a normal CPB without the use of any hemoadsorption system.
  Interventions: Device: Control

INTERVENTIONS:
Device: CytoSorb — The hemadsorption filter will be included in the CPB circuit between the oxygenator and the venous reservoir. After cardiac surgery, the use of the filter will be continued till 24 hours after the end of surgery.
  Arms: CytoSorb
Device: Control — No hemadsorption filter or other treatment will be included in the CPB circuit
  Arms: Control

SUMMARY:
Chronic kidney disease (CKD) is a risk factor for the development of cardiovascular disease, which increases the risk of death after cardiac surgery. High interleukin 6 (IL-6) blood levels is commonly observed in patients with CKD, and this is particularly high after cardiac surgery. High IL-6 levels are also associated with increased long-term mortality rate after cardiac surgery. To date, the use of ultrafiltration or endotoxin adsorption systems were not found to improve the clinical outcome, although able to reduce the inflammatory mediators concentrations. In the last years, a new extracorporeal hemadsorption filter (CytoSorb) has been developed for removal of inflammatory cytokines and it has been approved by the European Union. However, data lack about the impact on clinical outcome of the use of CytoSorb in patients with CKD undergoing cardiac surgery with cardio-pulmonary bypass (CPB). The investigators have therefore designed this pilot prospective randomized trial to evaluate the efficacy the intraoperative use of CytoSorb for cytokines removal to prevent the inflammatory response associated with the cardiac surgery and complications in patients with CKD.

ELIGIBILITY:
Inclusion Criteria:

* All consecutive adult patients (age >65 years) undergoing cardiac surgery with an anticipated CPB time duration longer than 60 minutes.
* Presence of CKD defined by a Glomerular Filtration Rate (eGFR) < 60 ml/min/1.73 m2.
* Consent to participate to the study

Exclusion Criteria:

* emergency surgery
* acute infective endocarditis
* systemic infectious diseases
* previous kidney transplant
* need for contrast enhancement during surgery
* immunosuppressive or long-term corticosteroid therapies
* participation to other investigations.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-11-15 (Estimated); Primary Completion 2021-11-01 (Estimated); Study Completion 2021-11-15 (Estimated)

PRIMARY OUTCOMES:
IL-6 concentration at ICU admission | At day 0 after surgery
  Investigators will assess the blood IL-6 concentrations between the two arms

SECONDARY OUTCOMES:
IL-6 concentration before cardiac surgery | At day 0 before the cardiac surgery
  Investigators will assess the blood IL-6 concentrations between the two arms
IL-6 concentration at the end of CardioPulmonary Bypass | At day 0 at the end of the CardioPulmonary Bypass
  Investigators will assess the blood IL-6 concentrations between the two arms
IL-6 concentration 2 hours after the end of CardioPulmonary Bypass | 2 hours after the end of CardioPulmonary Bypass
  Investigators will assess the blood IL-6 concentrations between the two arms
IL-6 concentration 48 hours after the end of CardioPulmonary Bypass | 48 hours after the end of CardioPulmonary Bypass
  Investigators will assess the blood IL-6 concentrations between the two arms
Renal function | daily up to day 15
  Investigators will assess the blood creatinine concentrations in the two arms
Myoglobin concentration | daily up to day 15
  Investigators will assess the blood myoglobin concentrations in the two arms
Haptoglobin concentration | daily up to day 15
  Investigators will assess the blood haptoglobin concentrations in the two arms
Liver transaminases concentration | daily up to day 15
  Investigators will measure the liver transaminases concentrations in the two arms to assess any liver injury
Osteopontin concentration | daily up to day 15
  Investigators will measure the osteopontin concentrations in the two arms to assess the inflammatory status
Free hemoglobin concentration | daily up to day 15
  Investigators will assess the free hemoglobin concentrations in the two arms

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Serraino, MD, Principal Investigator — Magna Graecia University
Locations (1):
- AOU Mater Domini, Catanzaro, CZ, Italy

IPD SHARING:
Plan to Share IPD: Yes
The full protocol, datasets used and analysed during the current study will be available on reasonable request after study publication
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: After scientific publication
Access Criteria: On reasonable request

REFERENCES:
- [Background] Tonelli M, Wiebe N, Culleton B, House A, Rabbat C, Fok M, McAlister F, Garg AX. Chronic kidney disease and mortality risk: a systematic review. J Am Soc Nephrol. 2006 Jul;17(7):2034-47. doi: 10.1681/ASN.2005101085. Epub 2006 May 31. PMID 16738019
- [Background] Penta de Peppo A, Nardi P, De Paulis R, Pellegrino A, Forlani S, Scafuri A, Chiariello L. Cardiac surgery in moderate to end-stage renal failure: analysis of risk factors. Ann Thorac Surg. 2002 Aug;74(2):378-83. doi: 10.1016/s0003-4975(02)03711-6. PMID 12173816
- [Background] Durmaz I, Buket S, Atay Y, Yagdi T, Ozbaran M, Boga M, Alat I, Guzelant A, Basarir S. Cardiac surgery with cardiopulmonary bypass in patients with chronic renal failure. J Thorac Cardiovasc Surg. 1999 Aug;118(2):306-15. doi: 10.1016/S0022-5223(99)70221-7. PMID 10425004
- [Background] Pecoits-Filho R, Heimburger O, Barany P, Suliman M, Fehrman-Ekholm I, Lindholm B, Stenvinkel P. Associations between circulating inflammatory markers and residual renal function in CRF patients. Am J Kidney Dis. 2003 Jun;41(6):1212-8. doi: 10.1016/s0272-6386(03)00353-6. PMID 12776273
- [Background] Takahashi T, Kubota M, Nakamura T, Ebihara I, Koide H. Interleukin-6 gene expression in peripheral blood mononuclear cells from patients undergoing hemodialysis or continuous ambulatory peritoneal dialysis. Ren Fail. 2000 May;22(3):345-54. doi: 10.1081/jdi-100100878. PMID 10843245
- [Background] Caglar K, Peng Y, Pupim LB, Flakoll PJ, Levenhagen D, Hakim RM, Ikizler TA. Inflammatory signals associated with hemodialysis. Kidney Int. 2002 Oct;62(4):1408-16. doi: 10.1111/j.1523-1755.2002.kid556.x. PMID 12234313
- [Background] Corral-Velez V, Lopez-Delgado JC, Betancur-Zambrano NL, Lopez-Sune N, Rojas-Lora M, Torrado H, Ballus J. The inflammatory response in cardiac surgery: an overview of the pathophysiology and clinical implications. Inflamm Allergy Drug Targets. 2015;13(6):367-70. doi: 10.2174/1871528114666150529120801. PMID 26021321
- [Background] de Amorim CG, Malbouisson LM, da Silva FC Jr, Fiorelli AI, Murakami CK, Carmona MJ. Leukocyte depletion during CPB: effects on inflammation and lung function. Inflammation. 2014 Feb;37(1):196-204. doi: 10.1007/s10753-013-9730-z. PMID 24092406
- [Background] Ilmakunnas M, Pesonen EJ, Ahonen J, Ramo J, Siitonen S, Repo H. Activation of neutrophils and monocytes by a leukocyte-depleting filter used throughout cardiopulmonary bypass. J Thorac Cardiovasc Surg. 2005 Apr;129(4):851-9. doi: 10.1016/j.jtcvs.2004.07.061. PMID 15821654
- [Background] Wiegele M, Krenn CG. Cytosorb in a patient with Legionella pneumonia-associated rhabdomyolysis: a case report. ASAIO J. 2015 May-Jun;61(3):e14-6. doi: 10.1097/MAT.0000000000000197. No abstract available. PMID 25635933
- [Background] Basu R, Pathak S, Goyal J, Chaudhry R, Goel RB, Barwal A. Use of a novel hemoadsorption device for cytokine removal as adjuvant therapy in a patient with septic shock with multi-organ dysfunction: A case study. Indian J Crit Care Med. 2014 Dec;18(12):822-4. doi: 10.4103/0972-5229.146321. PMID 25538418
- [Background] Hetz H, Berger R, Recknagel P, Steltzer H. Septic shock secondary to beta-hemolytic streptococcus-induced necrotizing fasciitis treated with a novel cytokine adsorption therapy. Int J Artif Organs. 2014 May;37(5):422-6. doi: 10.5301/ijao.5000315. Epub 2014 Apr 17. PMID 24811308
- [Background] Vercaemst L. Hemolysis in cardiac surgery patients undergoing cardiopulmonary bypass: a review in search of a treatment algorithm. J Extra Corpor Technol. 2008 Dec;40(4):257-67. PMID 19192755
- [Background] Kahles F, Findeisen HM, Bruemmer D. Osteopontin: A novel regulator at the cross roads of inflammation, obesity and diabetes. Mol Metab. 2014 Mar 22;3(4):384-93. doi: 10.1016/j.molmet.2014.03.004. eCollection 2014 Jul. PMID 24944898
- [Background] Baumann A, Buchwald D, Annecke T, Hellmich M, Zahn PK, Hohn A. RECCAS - REmoval of Cytokines during CArdiac Surgery: study protocol for a randomised controlled trial. Trials. 2016 Mar 12;17(1):137. doi: 10.1186/s13063-016-1265-9. PMID 26971164